CLINICAL TRIAL: NCT05389839
Title: Application of Intelligent Insulin Dose Calculation Software in Patients With Insulin Therapy：A Randomized Controlled Intervention Trial
Brief Title: Insulin Dose Calculation Software in Insulin Therapy
Acronym: IDCST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: xiaolong zhao (Other)
Responsible Party: Sponsor-Investigator, xiaolong zhao, director, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21Y11904700
Record Dates: First submitted 2021-10-25; First posted 2022-05-25 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Time in Range; Artificial Intelligence; Insulin Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wechat program guidance group (Experimental): Wechat program guidance group using insulin dose calculator
  Interventions: Device: Wechat program
- clinical experience treatment group (Active Comparator): clinical experience treatment group using physician experience
  Interventions: Device: Wechat program

INTERVENTIONS:
Device: Wechat program — The experimental group used wechat program to calculate insulin dose to guide insulin treatment .

SUMMARY:
Insulin therapy is the mainstream glucose-lowering program for hospital glucose management. Intelligent insulin dose calculation software based on fingertip glucose monitoring is born in response to the situation. A new generation of continuous blood glucose monitoring technology compared with traditional monitoring technology provides more abundant blood sugar change information.The development of the continuous glucose monitoring technology espcially in blood sugar change trend arrow information, the intelligent insulin dose adjustment sequence based on WeChat program is developed. We plan to carry out a randomized controlled study on patients receiving insulin therapy, in which the insulin dose is adjusted according to the information of four blood glucose monitoring points (before meals and before bed), and randomly divided into two groups, one group is adjusted according to the experience of clinicians, the other group is adjusted according to Wechat program, and glucose monitoring is continued for 1 week. bBood glucose control index of TIR , and the incidence of hypoglycemia and hyperglycemia, hospitalization days and cost was observed. This study ihas great clinical value.

DETAILED DESCRIPTION:
The problems related to blood glucose in non-endocrine departments are becoming more and more serious.Glucose control level is closely related to the prognosis and cost of inpatients. Insulin therapy is the mainstream glucose-lowering program for hospital glucose management. Intelligent insulin dose calculation software based on fingertip glucose monitoring is born in response to the situation. A new generation of continuous blood glucose monitoring technology compared with traditional monitoring technology provides more abundant blood sugar change information.The development of the continuous glucose monitoring technology espcially in blood sugar change trend arrow information, the intelligent insulin dose adjustment sequence based on WeChat program is developed. We plan to carry out a randomized controlled study on patients receiving insulin therapy, in which the insulin dose is adjusted according to the information of four blood glucose monitoring points (before meals and before bed), and randomly divided into two groups, one group is adjusted according to the experience of clinicians, the other group is adjusted according to Wechat program, and glucose monitoring is continued for 1 week. bBood glucose control index of TIR , and the incidence of hypoglycemia and hyperglycemia, hospitalization days and cost was observed. This study ihas great clinical value.

ELIGIBILITY:
Inclusion Criteria:

* 1. Non-endocrine departments;
* 2. Age 18-70;
* 3. Currently using intensive insulin therapy with basic meals;
* 4. Belong to type 1 or Type 2 diabetes
* 5. Hospitalized patients 6. Regular meals

Exclusion Criteria:

* 1. Unwilling to participate or unable to cooperate.
* 2. Myocardial infarction or cardiovascular and cerebrovascular events in the last 3 months;
* 3. Glomerular filtration rate < 45 ml/min / 1.73 m2;
* 4. Other serious concomitant diseases;
* 5. Liver function transaminase is 2 times higher than the upper limit of normal range;
* 6. Use of oral hypoglycemic drugs other than metformin
* 7. Asymptomatic hypoglycemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Subjects in both groups targeted blood glucose range (TIR) time or ratio. | one week
  Subjects in both groups targeted blood glucose range (TIR) time or ratio.

SECONDARY OUTCOMES:
Mean blood glucose | one week
  Mean blood glucose
above target blood glucose range (TAR) for time or ratio, | one week
  above target blood glucose range (TAR) for time or ratio,
below target blood glucose range (TBR) for time or Proportion | one week
  below target blood glucose range (TBR) for time or Proportion
insulin dose | one week
  insulin dose
hospitalization cost | one week
  hospitalization cost
hospitalization length of stay | one week
  hospitalization length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Zhao, PhD, Study Chair — Shanghai Public Health Clinical Center
Locations (1):
- Xiaolong Zhao, Shanghai, Shanghai Municipality, China